CLINICAL TRIAL: NCT05990218
Title: Efficacy of Artificial Intelligence in the Detection of Right Sided Colonic Polyp in Operators with Different Endoscopic Experience: a Randomized Control Trial
Brief Title: Artificial Intelligence in the Detection of Right Sided Colonic Polyp in Different Operator Experience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 031/2566
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Colon Polyp
Keywords: colon polyp; artificial intellegence; colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Patients randomized to 4 arms: control with experienced operator, control with beginner operator, AI with experienced operator, AI with beginner operator
Who Masked: Participant
Masking Description: The patients were masked from being randomized to operator and endoscopic method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control, experienced (Active Comparator): Patients received colonoscopy with double insertion of right sided colon under white light by experienced endoscopist
  Interventions: Device: control
- control, beginner (Active Comparator): Patients received colonoscopy with double insertion of right sided colon under white light by beginner endoscopist
  Interventions: Device: control
- AI, experience (Experimental): Patients received colonoscopy with double insertion of right sided colon under AI by experienced endoscopist
  Interventions: Device: Artificial intellegence. CADe syste,
- AI, beginner (Experimental): Patients received colonoscopy with double insertion of right sided colon under AI by beginner endoscopist
  Interventions: Device: Artificial intellegence. CADe syste,

INTERVENTIONS:
Device: Artificial intellegence. CADe syste, — The patient received endoscopy under CADe system for polyp detection during second endoscopic withdrawal.
  Arms: AI, beginner; AI, experience
Device: control — The patient received endoscopy under conventional white light for polyp detection during second endoscopic withdrawal.
  Arms: control, beginner; control, experienced

SUMMARY:
Colonoscopy is the gold standard modality for the detection of colonic polyp. However, miss polyp occurs especially in right sided colon. Artificial intelligence (AI) is one of the modality to improve polyp detection but the benefit of AI in operators with different endoscopic experience is still limited. This study aimed to evaluate the efficacy of AI in the detection of right sided colonic polyp in operators with different endoscopic experience by using double insertion of right side colon, back-to-back basis.

ELIGIBILITY:
Inclusion Criteria:

* participants age 40-80 years

Exclusion Criteria:

* History of colonic surgery (except appendectomy)
* Lower gastrointestinal bleeding
* unstable vital sign during endoscopy of pregnancy
* history of inflammatory bowel disease, polyposis syndrome, colon cancer, colonic stricture, abnormal coaglulation, organ failure

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
polyp detection rate | during endoscopy
  the number of polyp detected during endoscopy

SECONDARY OUTCOMES:
type of polyp | during endoscopy
  the type of polyp detected during endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamba S, Tamai N, Saitoh I, Matsui H, Horiuchi H, Kobayashi M, Sakamoto T, Ego M, Fukuda A, Tonouchi A, Shimahara Y, Nishikawa M, Nishino H, Saito Y, Sumiyama K. Reducing adenoma miss rate of colonoscopy assisted by artificial intelligence: a multicenter randomized controlled trial. J Gastroenterol. 2021 Aug;56(8):746-757. doi: 10.1007/s00535-021-01808-w. Epub 2021 Jul 3. PMID 34218329